CLINICAL TRIAL: NCT02573506
Title: A Prospective Phase Ⅱ Study of Split-course Chemoradiotherapy For Locally Advanced None-small Cell Lung Cancer
Brief Title: Study of Split-course Chemoradiotherapy For Locally Advanced None-small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hui Liu, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GASTO1011
Record Dates: First submitted 2015-09-19; First posted 2015-10-09 (Estimated); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Non-small cell lung cancer; Split-course Chemoradiotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- split-course radiotherapy (Experimental): The radiotherapy is delivered using simultaneous integrated boost (SIB)-IMRT. Patients are irradiation at a palliative dose in the initial course: 51Gy/17f to PTV-GTV. The disease is re-evaluated three weeks after the end of the initial course using CT. The patient without disease progression according to the RECIST criteria and had a recovery of lung function should get the additional boost. In the second course, the tumor is repositioned and scanned. The residual tumor is then treated with the second course of radiotherapy. A dose of 15-18 Gy/5-6f is delivered to the residue tumor. Concurrent chemotherapy consists of weekly docetaxel(25mg/㎡) and nedaplatin(25mg/㎡), each of 1 day's duration.
  Interventions: Radiation: split-course radiotherapy; Drug: Concurrent chemotherapy

INTERVENTIONS:
Radiation: split-course radiotherapy — Patients are irradiation at a palliative dose in the initial course: 51Gy/17f to PTV-GTV. The disease is re-evaluated three weeks after the end of the initial course using CT. The patient without disease progression according to the RECIST criteria and had a recovery of lung function should get the additional boost. In the second course, the tumor is repositioned and scanned. The residual tumor is then treated with the second course of radiotherapy. A dose of 15-18 Gy/5-6f is delivered to the residue tumor.
Drug: Concurrent chemotherapy — Concurrent chemotherapy consists of weekly docetaxel(25mg/㎡) and nedaplatin(25mg/㎡), each of 1 day's duration.

SUMMARY:
This Phase II study is to determine the efficacy of split-course irradiation with concurrent chemotherapy in locally advanced none-small cell lung cancer patients.

DETAILED DESCRIPTION:
This Phase II study is to determine the efficacy of split-course chemoradiotherapy(CCRT) in locally advanced non-small cell lung cancer.

Patients receive four cycles of weekly docetaxel(25mg/㎡) and nedaplatin(25mg/㎡), each of 1 day's duration, combined with split-course thoracic radiotherapy of 51 Gy/17 fractions and 15-18 Gy/5-6 fractions administered in the first and second courses, respectively, with about one-month break. The primary endpoint is progression-free survival, which is calculated from the start of RT to the first identification of disease progression or death. Progression-free survival will be calculated using the Kaplan-Meier method. Toxicities will be graded according to CTCAE V.4.0.

ELIGIBILITY:
Inclusion Criteria:

* Pathologic confirmation of NSCLC.
* Patients have measurable or evaluable lesions based on the Response Evaluation Criteria in Solid Tumors (RECIST) criteria.
* Unresectable phase IIIA(N2) and IIIB lung cancer confirmed by PET/CT, CT or MRI.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
* Previously treated with chemotherapy or treatment-naive
* No previous chest radiotherapy, immunotherapy or biotherapy
* Hemoglobin≥10 mg/dL, platelet≥100000/μL,absolute neutrophil count ≥1500/μL
* Serum creatinine ≤1.25 times the upper normal limit(UNL), or creatinine clearance≥60 ml/min
* Bilirubin ≤1.5 times UNL, AST（SGOT）≤2.5 times UNL ,ALT（SGPT）≤2.5 times UNL,alkaline phosphatase ≤5 times UNL
* FEV1 >0.8 L
* CB6 within normal limits
* patients and their family signed the informed consents

Exclusion Criteria:

* Previous or recent another malignancy, except nonmelanoma skin cancer or cervical cancer in situ
* Contraindication for chemotherapy
* Malignant pleural or pericardial effusion.
* Women in pregnancy, lactation period, or no pregnancy test 14 days before the first dose
* Women who has the probability of pregnancy without contraception
* Tendency of hemorrhage
* In other clinical trials within 30 days
* Addicted in drugs or alcohol, AIDS patients
* Uncontrollable seizure or psychotic patients without self-control ability
* Severe allergy or idiosyncrasy
* Not suitable for this study judged by researchers

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2020-03 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
progression-free survival | 3 years

SECONDARY OUTCOMES:
Overall Survival | 3 years
Response Rate | 3 years
rate of grade 3-4 radiation esophagitis | 1 year
rate of grade 3-4 radiation pneumonitis | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Hui Liu, Doctor, Principal Investigator — Sun yat-sen universtiy cancer center
Locations (1):
- Hui Liu, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Steel GG, Hill RP, Peckham MJ. Combined radiotherapy--chemotherapy of Lewis lung carcinoma. Int J Radiat Oncol Biol Phys. 1978 Jan-Feb;4(1-2):49-52. doi: 10.1016/0360-3016(78)90114-1. No abstract available. PMID 632147
- [Background] Chemotherapy in non-small cell lung cancer: a meta-analysis using updated data on individual patients from 52 randomised clinical trials. Non-small Cell Lung Cancer Collaborative Group. BMJ. 1995 Oct 7;311(7010):899-909. PMID 7580546
- [Background] Marino P, Preatoni A, Cantoni A. Randomized trials of radiotherapy alone versus combined chemotherapy and radiotherapy in stages IIIa and IIIb nonsmall cell lung cancer. A meta-analysis. Cancer. 1995 Aug 15;76(4):593-601. doi: 10.1002/1097-0142(19950815)76:43.0.co;2-n. PMID 8625152
- [Background] Pritchard RS, Anthony SP. Chemotherapy plus radiotherapy compared with radiotherapy alone in the treatment of locally advanced, unresectable, non-small-cell lung cancer. A meta-analysis. Ann Intern Med. 1996 Nov 1;125(9):723-9. doi: 10.7326/0003-4819-125-9-199611010-00003. PMID 8929005
- [Background] Kubota K, Furuse K, Kawahara M, Kodama N, Yamamoto M, Ogawara M, Negoro S, Masuda N, Takada M, Matsui K, et al. Role of radiotherapy in combined modality treatment of locally advanced non-small-cell lung cancer. J Clin Oncol. 1994 Aug;12(8):1547-52. doi: 10.1200/JCO.1994.12.8.1547. PMID 8040666
- [Background] Clinical practice guidelines for the treatment of unresectable non-small-cell lung cancer. Adopted on May 16, 1997 by the American Society of Clinical Oncology. J Clin Oncol. 1997 Aug;15(8):2996-3018. doi: 10.1200/JCO.1997.15.8.2996. PMID 9256144
- [Background] Curran WJ, Scott C, Langer C, et al. Phase III comoarision of sequential vs concurrent chemoradiation therapy for patients with unresectable stage III non-small cell lung cancer: initial report of RTOG 9410. Proc Am Soc Clin Oncol, 2000, 19: 484a
- [Background] Furuse K, Fukuoka M, Kawahara M, Nishikawa H, Takada Y, Kudoh S, Katagami N, Ariyoshi Y. Phase III study of concurrent versus sequential thoracic radiotherapy in combination with mitomycin, vindesine, and cisplatin in unresectable stage III non-small-cell lung cancer. J Clin Oncol. 1999 Sep;17(9):2692-9. doi: 10.1200/JCO.1999.17.9.2692. PMID 10561343
- [Background] Auperin A, Le Pechoux C, Rolland E, Curran WJ, Furuse K, Fournel P, Belderbos J, Clamon G, Ulutin HC, Paulus R, Yamanaka T, Bozonnat MC, Uitterhoeve A, Wang X, Stewart L, Arriagada R, Burdett S, Pignon JP. Meta-analysis of concomitant versus sequential radiochemotherapy in locally advanced non-small-cell lung cancer. J Clin Oncol. 2010 May 1;28(13):2181-90. doi: 10.1200/JCO.2009.26.2543. Epub 2010 Mar 29. PMID 20351327
- [Background] Pfister DG, Johnson DH, Azzoli CG, Sause W, Smith TJ, Baker S Jr, Olak J, Stover D, Strawn JR, Turrisi AT, Somerfield MR; American Society of Clinical Oncology. American Society of Clinical Oncology treatment of unresectable non-small-cell lung cancer guideline: update 2003. J Clin Oncol. 2004 Jan 15;22(2):330-53. doi: 10.1200/JCO.2004.09.053. Epub 2003 Dec 22. No abstract available. PMID 14691125
- [Background] Ardizzoni A, Tiseo M, Boni L et al. CISCA (cis-platin vs. carboplatin) meta-analysis: an individual patient data meta-analysis comparing cisplatin versus carboplatin-based chemotherapy in first-line treatment of advanced non-small cell lung cancer (NSCLC) [Abstract 7011]. Proc AmSoc Clin Oncol 2006;24:366S.
- [Background] Blackstock AW, Socinski MA, Bogart J, et al; Cancer and Leukemia Group B. Induction plus concurrent chemotherapy with high-dose (74 Gy) 3-dimensional (3-D) thoracic radiotherapy in stage III non-small cell lung cancer. Preliminary report of Cancer and Leukemia Group B (CALGB) 30105. Proc Am Soc Clin Oncol 2006;24(18S):Abstr 7042
- [Background] Lee CB, Socinski A, Lin L, et al. High-dose 3D chemoradiotherapy in stage III non-small cell lung cancer (NSCLC) at the University of North Carolina: long-term follow up and late complications. Proc Am Soc Clin Oncol 2006;24(18S):Abstr 7145.
- [Background] Kong FM, Ten Haken RK, Schipper MJ, Sullivan MA, Chen M, Lopez C, Kalemkerian GP, Hayman JA. High-dose radiation improved local tumor control and overall survival in patients with inoperable/unresectable non-small-cell lung cancer: long-term results of a radiation dose escalation study. Int J Radiat Oncol Biol Phys. 2005 Oct 1;63(2):324-33. doi: 10.1016/j.ijrobp.2005.02.010. PMID 16168827
- [Background] Schild SE, McGinnis WL, Graham D, Hillman S, Fitch TR, Northfelt D, Garces YI, Shahidi H, Tschetter LK, Schaefer PL, Adjei A, Jett J. Results of a Phase I trial of concurrent chemotherapy and escalating doses of radiation for unresectable non-small-cell lung cancer. Int J Radiat Oncol Biol Phys. 2006 Jul 15;65(4):1106-11. doi: 10.1016/j.ijrobp.2006.02.046. Epub 2006 May 26. PMID 16730134
- [Background] Bradley JD, Paulus R, Komaki R, Masters G, Blumenschein G, Schild S, Bogart J, Hu C, Forster K, Magliocco A, Kavadi V, Garces YI, Narayan S, Iyengar P, Robinson C, Wynn RB, Koprowski C, Meng J, Beitler J, Gaur R, Curran W Jr, Choy H. Standard-dose versus high-dose conformal radiotherapy with concurrent and consolidation carboplatin plus paclitaxel with or without cetuximab for patients with stage IIIA or IIIB non-small-cell lung cancer (RTOG 0617): a randomised, two-by-two factorial phase 3 study. Lancet Oncol. 2015 Feb;16(2):187-99. doi: 10.1016/S1470-2045(14)71207-0. Epub 2015 Jan 16. PMID 25601342
- [Background] Spoelstra FO, Pantarotto JR, van Sornsen de Koste JR, Slotman BJ, Senan S. Role of adaptive radiotherapy during concomitant chemoradiotherapy for lung cancer: analysis of data from a prospective clinical trial. Int J Radiat Oncol Biol Phys. 2009 Nov 15;75(4):1092-7. doi: 10.1016/j.ijrobp.2008.12.027. Epub 2009 Mar 26. PMID 19327915
- [Background] Gielda BT, Marsh JC, Zusag TW, Faber LP, Liptay M, Basu S, Warren WH, Fidler MJ, Batus M, Abrams RA, Bonomi P. Split-course chemoradiotherapy for locally advanced non-small cell lung cancer: a single-institution experience of 144 patients. J Thorac Oncol. 2011 Jun;6(6):1079-86. doi: 10.1097/JTO.0b013e3182199a7c. PMID 21532501
- [Background] Belani CP, Choy H, Bonomi P, Scott C, Travis P, Haluschak J, Curran WJ Jr. Combined chemoradiotherapy regimens of paclitaxel and carboplatin for locally advanced non-small-cell lung cancer: a randomized phase II locally advanced multi-modality protocol. J Clin Oncol. 2005 Sep 1;23(25):5883-91. doi: 10.1200/JCO.2005.55.405. Epub 2005 Aug 8. PMID 16087941
- [Background] Curran W, Scott C, Langer C, et al. Phase III comparison of sequential vs concurrent chemoradiotherapy for patients (pts) with unresected stage III non-small cell lung cancer (NSCLC): report of Radiation Therapy Oncology Group (RTOG) 9410. Proc Am Soc Clin Oncol 2003;22:Abstr 2499.
- [Background] Albain KS, Swann RS, Rusch VW, Turrisi AT 3rd, Shepherd FA, Smith C, Chen Y, Livingston RB, Feins RH, Gandara DR, Fry WA, Darling G, Johnson DH, Green MR, Miller RC, Ley J, Sause WT, Cox JD. Radiotherapy plus chemotherapy with or without surgical resection for stage III non-small-cell lung cancer: a phase III randomised controlled trial. Lancet. 2009 Aug 1;374(9687):379-86. doi: 10.1016/S0140-6736(09)60737-6. Epub 2009 Jul 24. PMID 19632716
- [Background] Vokes EE, Herndon JE 2nd, Kelley MJ, Cicchetti MG, Ramnath N, Neill H, Atkins JN, Watson DM, Akerley W, Green MR; Cancer and Leukemia Group B. Induction chemotherapy followed by chemoradiotherapy compared with chemoradiotherapy alone for regionally advanced unresectable stage III Non-small-cell lung cancer: Cancer and Leukemia Group B. J Clin Oncol. 2007 May 1;25(13):1698-704. doi: 10.1200/JCO.2006.07.3569. Epub 2007 Apr 2. PMID 17404369
- [Background] Hanna N, Neubauer M, Yiannoutsos C, McGarry R, Arseneau J, Ansari R, Reynolds C, Govindan R, Melnyk A, Fisher W, Richards D, Bruetman D, Anderson T, Chowhan N, Nattam S, Mantravadi P, Johnson C, Breen T, White A, Einhorn L; Hoosier Oncology Group; US Oncology. Phase III study of cisplatin, etoposide, and concurrent chest radiation with or without consolidation docetaxel in patients with inoperable stage III non-small-cell lung cancer: the Hoosier Oncology Group and U.S. Oncology. J Clin Oncol. 2008 Dec 10;26(35):5755-60. doi: 10.1200/JCO.2008.17.7840. Epub 2008 Nov 10. PMID 19001323
- [Background] Segawa Y, Kiura K, Takigawa N, Kamei H, Harita S, Hiraki S, Watanabe Y, Sugimoto K, Shibayama T, Yonei T, Ueoka H, Takemoto M, Kanazawa S, Takata I, Nogami N, Hotta K, Hiraki A, Tabata M, Matsuo K, Tanimoto M. Phase III trial comparing docetaxel and cisplatin combination chemotherapy with mitomycin, vindesine, and cisplatin combination chemotherapy with concurrent thoracic radiotherapy in locally advanced non-small-cell lung cancer: OLCSG 0007. J Clin Oncol. 2010 Jul 10;28(20):3299-306. doi: 10.1200/JCO.2009.24.7577. Epub 2010 Jun 7. PMID 20530281
- [Background] Davies AM, Chansky K, Lau DH, Leigh BR, Gaspar LE, Weiss GR, Wozniak AJ, Crowley JJ, Gandara DR; SWOG S9712. Phase II study of consolidation paclitaxel after concurrent chemoradiation in poor-risk stage III non-small-cell lung cancer: SWOG S9712. J Clin Oncol. 2006 Nov 20;24(33):5242-6. doi: 10.1200/JCO.2006.07.0268. PMID 17114656
- [Background] Fu KK, Pajak TF, Trotti A, Jones CU, Spencer SA, Phillips TL, Garden AS, Ridge JA, Cooper JS, Ang KK. A Radiation Therapy Oncology Group (RTOG) phase III randomized study to compare hyperfractionation and two variants of accelerated fractionation to standard fractionation radiotherapy for head and neck squamous cell carcinomas: first report of RTOG 9003. Int J Radiat Oncol Biol Phys. 2000 Aug 1;48(1):7-16. doi: 10.1016/s0360-3016(00)00663-5. PMID 10924966
- [Background] Saunders M, Dische S, Barrett A, Harvey A, Griffiths G, Palmar M. Continuous, hyperfractionated, accelerated radiotherapy (CHART) versus conventional radiotherapy in non-small cell lung cancer: mature data from the randomised multicentre trial. CHART Steering committee. Radiother Oncol. 1999 Aug;52(2):137-48. doi: 10.1016/s0167-8140(99)00087-0. PMID 10577699
- [Background] Petereit DG, Sarkaria JN, Chappell R, Fowler JF, Hartmann TJ, Kinsella TJ, Stitt JA, Thomadsen BR, Buchler DA. The adverse effect of treatment prolongation in cervical carcinoma. Int J Radiat Oncol Biol Phys. 1995 Jul 30;32(5):1301-7. doi: 10.1016/0360-3016(94)00635-X. PMID 7635769
- [Background] Begg AC, Hofland I, Van Glabekke M, et al. Predictive value of potential doubling time for radiotherapy of head and neck tumor pa- tients: results from the EORTC cooperative trial 22851. Semin Radiat Oncol 1992;2:22-25
- [Background] Kim YS, Choi EK, Lee JS et al. Consolidation chemotherapy with monthly Paclitaxel and Cisplatin (PC) or observation after concurrent chemoradiotherapy for locally advanced non-small cell lung cancer (NSCLS): randomized phase II study. J Thorac Oncol 2007; 2:449s.
- [Background] Huber R, M, Engel-Riedel W, Kollmeier J et al. GILT study: oral vinorel- bine (NVBo) and cisplatin (P) with concomitant radiotherapy (RT) fol- lowed by either consolidation (C) with NVBo plus P plus best supportive care (BSC) or BSC alone in stage (st) III non-small cell lung cancer (NSCLC): final results of a phase (ph) III study. J Clin Oncol 2012;30: 452s (suppl, abstr 7001).
- [Background] Ahn JS, Ahn YC, Kim JH, Lee CG, Cho EK, Lee KC, Chen M, Kim DW, Kim HK, Min YJ, Kang JH, Choi JH, Kim SW, Zhu G, Wu YL, Kim SR, Lee KH, Song HS, Choi YL, Sun JM, Jung SH, Ahn MJ, Park K. Multinational Randomized Phase III Trial With or Without Consolidation Chemotherapy Using Docetaxel and Cisplatin After Concurrent Chemoradiation in Inoperable Stage III Non-Small-Cell Lung Cancer: KCSG-LU05-04. J Clin Oncol. 2015 Aug 20;33(24):2660-6. doi: 10.1200/JCO.2014.60.0130. Epub 2015 Jul 6. PMID 26150444
- [Background] Tsujino K, Kurata T, Yamamoto S, Kawaguchi T, Kubo A, Isa S, Hasegawa Y, Ou SH, Takada M, Ando M. Is consolidation chemotherapy after concurrent chemo-radiotherapy beneficial for patients with locally advanced non-small-cell lung cancer? A pooled analysis of the literature. J Thorac Oncol. 2013 Sep;8(9):1181-9. doi: 10.1097/JTO.0b013e3182988348. PMID 23883782
- [Derived] Qiu B, Xi Y, Liu F, Li Y, Xie X, Guo J, Guo S, Wu Y, Wu L, Liang T, Ding Y, Zhang J, Wu Q, Liu H. Gut Microbiome Is Associated With the Response to Chemoradiotherapy in Patients With Non-small Cell Lung Cancer. Int J Radiat Oncol Biol Phys. 2023 Feb 1;115(2):407-418. doi: 10.1016/j.ijrobp.2022.07.032. Epub 2022 Jul 26. PMID 35905860